CLINICAL TRIAL: NCT00704626
Title: CCRC: Serum Auto-Antibodies in Neurological Disease
Brief Title: Serum Auto-Antibodies in Neurological Diseases
Acronym: SAA
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 215828
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Myasthenia Gravis; Transverse Myelitis
Keywords: Multiple Sclerosis; Autoimmune disease; Inflammatory disease; Myasthenia Gravis; Transverse Myelitis
MeSH Terms: conditions — Multiple Sclerosis; Myasthenia Gravis; Myelitis, Transverse; Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5cc of serum will be obtained from patients with multiple sclerosis and other autoimmune and inflammatory diseases of the nervous system. Samples may be processed immediately or at a later time. Samples will be stored frozen in the freezer located in the Neuroscience building at Research Park in Davis, CA. Samples are identified with initials only.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects with multiple sclerosis and other autoimmune and inflammatory disease of the nervous system
  Interventions: Other: Blood Draw; Other: Cheek swab

INTERVENTIONS:
Other: Blood Draw — A 5cc sample of serum will be drawn from each subject. Only one blood draw is required, but up to 8 additional blood draws can be obtained.
Other: Cheek swab — A swab will be swished around the inside of the mouth to collect mouth (buccal) cells. This will be done with each blood draw.
  Other Names: Buccal swab

SUMMARY:
Under normal conditions our immune system protects us against infections and tumors. The immune system does this by recognizing that the infecting organism or the tumor is foreign to the body and attacking it. One way the immune system attacks a foreign target is by making proteins called antibodies that bind to the target. Sometimes, for reasons we poorly understand, the immune system wrongly identifies part of our own body as being foreign and attacks it. This can result in disease such as some forms of diabetes and thyroid disease, as well as some neurological diseases. In this study, one tablespoon of blood will be removed from each subject and tested to see if the immune system is making antibodies against components of the nerves and muscles. We also hope to learn if these antibodies contribute to the development or worsening of illnesses of the nervous system. Only one blood draw is required, but subjects may be asked to give up to 8 additional blood samples to see if the level of antibodies changes over time. Any additional blood draws would be performed at regularly scheduled clinic visits. There would be at least 3 months between blood draws over a period of up to 3 years, if requested by the physician.

Depending on your diagnosis, the physician may also request the collection of mouth (buccal) cells. This takes about one minute and is painless. The cells are collected by swishing a swab around your mouth. This cheek swab would be done with each blood draw.

Please note that this study is conducted ONLY at UC Davis and that all participants must be seen in our clinic located in Sacramento, CA. Results of the testing performed in this study are not given to the participants. This study is not intended to treat or diagnose any condition.

DETAILED DESCRIPTION:
The purposes of the study are to determine the frequency of auto-antibodies to 1) heat shock proteins and 2) to other molecules including cytoskeletal proteins such as rapsyn in diseases of the nervous system.

5cc of serum will be obtained from patients with multiple sclerosis and other autoimmune and inflammatory diseases of the nervous system including myasthenia gravis and transverse myelitis and from patients with other neurological diseases. Standard methodology to assure safe handling of serum will be used. Diluted serum will be tested for specific reactivity with heat shock proteins (Sigma Chemical Co., St. Louis, MO) as well as with other antigens in a standard ELISA as well as immunoblot.

Buccal swab will also be obtained in conjunction with each blood draw. Rapsyn and other cytoskeletal proteins will be extracted from Torpedo californica electric organ by means of differential centrifugation followed by alkali extraction. For the ELISA, a standard titration curve will be obtained for a positive control serum as previously determined. Negative control sera will be obtained from individuals with other degenerative neurological diseases. Titers of test serum will be determined as the dilution that generates a positive result that is two standard deviations from the mean of the background. Positive ELISA results will be confirmed by immunoblot. Patients may be tested at one time point only. If the serum is positive for specific antibody binding, additional serum samples may be obtained and retested up to 8 more times approximately 3 months apart. Correlation with severity of clinical findings and specific antibody titer will be made. Severity of clinical findings will be determined by the neurological exam done by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of multiple sclerosis, myasthenia gravis, or other autoimmune or inflammatory neurological disease

Exclusion Criteria:

* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older with multiple sclerosis, myasthenia gravis and other autoimmune or inflammatory neurological illnesses will be selected for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2002-01; Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
If the serum is positive for specific antibody binding, additional serum samples may be obtained and retested up to 8 more times approximately 3 months apart. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Richman, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-antibodies-in-the-blood-in-patients-with-auto-immune-neurological-diseases-662406/